CLINICAL TRIAL: NCT07034456
Title: Possible Mechanisms of Action of Magnetic Tape Through Its Application on the Epidermis
Brief Title: Sensory and Vascular Effects of Kinesio and Magnetic Tape in Healthy Subjects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Patricia Beltra Lopez (Other)
Collaborators: Miguel Delicado Miralles (Unknown); Gustavo Adolfo Sarriá (Unknown); Enrique Velasco Serna (Unknown)
Responsible Party: Sponsor-Investigator, Patricia Beltra Lopez, BSc in Physiotherapy. MSc. PhD Candidate in Health Sciences. COFCV Registration No.: 6563, Clinica Francisco Ortega Rehabilitacion Avanzada SL
Organization: Clinica Francisco Ortega Rehabilitacion Avanzada SL (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Magnetic Tape/2025
Record Dates: First submitted 2025-06-11; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: Magnetic Tape; Cutaneous Stimulation; Somatosensory System; Blood Flow

STUDY DESIGN:
Intervention Model Description: A Clinical trial crossover design. Each participant will receive all four conditions combining two types of tape (magnetic vs. placebo) and two types of cream (anesthetic vs. moisturizing), in randomized order with one-week washout periods between session. This design is similar to 2x2 factorial, but with a repeated measures.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo Tape with Moisturizing Cream (Crossover) (Sham Comparator): Participants will receive Placebo Tape with moisturizing cream
  Each condition will be applied in a separate session with a one-week washout period. All participants complete every condition in randomized order.
  Interventions: Device: Control KinesioTape; Device: Moisturizing Cream (control)
- Magnetic Tape with moisturizing cream (Experimental): Participants will receive Magnetic Tape with moisturizing cream
  Each condition will be applied in a separate session with a one-week washout period. All participants complete every condition in randomized order.
  Interventions: Device: Tape with mangetic particles; Device: Moisturizing Cream (control)
- Magnetic Tape with anaesthetic cream (Experimental): Participants will receive Magnetic Tape with anaesthetic cream Each condition will be applied in a separate session with a one-week washout period. All participants complete every condition in randomized order.
  Interventions: Device: Tape with mangetic particles; Drug: Topical Anesthetic Cream
- Placebo Tape with Anesthetic Cream (Placebo Comparator): Participants will receive Placebo Tape with Anesthetic cream Each condition will be applied in a separate session with a one-week washout period. All participants complete every condition in randomized order.
  Interventions: Drug: Topical Anesthetic Cream; Device: Control KinesioTape

INTERVENTIONS:
Device: Tape with mangetic particles — An elastic adhesive tape containing magnetic particles, designed to be applied directly to the skin. In this study, the tape is applied to the lumbar region. The tape remains in place during standardized sensory and vascular measurements
  Arms: Magnetic Tape with anaesthetic cream; Magnetic Tape with moisturizing cream
Drug: Topical Anesthetic Cream — EMLA®, a topical anesthetic cream containing lidocaine and prilocaine, will be applied under occlusion prior to tape application during 30 minutes with the aim of anesthetize the cutaneous sensory receptors
  Arms: Magnetic Tape with anaesthetic cream; Placebo Tape with Anesthetic Cream
Device: Control KinesioTape — An elastic adhesive tape, designed to be applied directly to the skin. In this study, the tape is applied to the lumbar region. This tape does not content magnetic particles, thus is used as a comparator. The tape remains in place during standardized sensory and vascular measurements
  Arms: Placebo Tape with Anesthetic Cream; Placebo Tape with Moisturizing Cream (Crossover)
Device: Moisturizing Cream (control) — A neutral moisturizing cream (control) will be applied under occlusion prior to tape application during 30 minutes. The application will be blind and use as a placebo vs the anesthetic cream.
  Arms: Magnetic Tape with moisturizing cream; Placebo Tape with Moisturizing Cream (Crossover)

SUMMARY:
This study aims to evaluate the effects of a tape with magnetic particles versus a control kinesiotape on the skin's sensory and vascular responses in healthy volunteers. The tape is an elastic adhesive strip containing magnetic particles that may modulate sensory nerve endings. The hypothesis is that this magnetic tape can reduce pain and mechanical sensitivity and blood flow in the application area by stimulating cutaneous receptors.

Thirty healthy participants will receive four different combinations of two types of tapes (magnetic vs. placebo) and two creams (anesthetic vs. moisturizing), applied to the lower back in a randomized crossover design. Sensory thresholds and blood flow will be measured at three body regions: close to the application site (lower back), a segmentally related area (posterior thigh), and an unrelated distant site (forearm). Measurements will include pressure pain threshold, mechanical sensitivity, and tactile detection, using standardized tools and Doppler ultrasound

The study will help determine whether the effects of magnetic tape are local or systemic, whether they depend on skin receptor activation, and whether they can be blocked by topical anesthesia

DETAILED DESCRIPTION:
This randomized, single-blind, crossover clinical trial investigates the sensory and vascular effects of an elastic adhesive tape containing magnetic particles (Magnetic Tape®) when applied to the skin of healthy volunteers. The study employs a 2x2 factorial design, combining two types of tape (magnetic vs. placebo) and two types of topical cream (anesthetic vs. moisturizing), applied in four different sessions with a one-week washout between conditions. Each participant receives all four combinations in a randomized order

The main hypothesis is that magnetic tape may induce local sensory and vascular changes through the activation of cutaneous sensory afferents. A secondary hypothesis is that these effects may be diminished or abolished by topical anesthetic application, indicating a dependence on superficial nerve activation. A third hypothesis is that any effects will be limited to the dermatome of application, without spreading to distant or segmentally unrelated areas

Sensory testing includes pressure pain threshold (PPT), mechanical pain sensitivity (using numeric rating scale), and tactile detection threshold (using von Frey filaments). These assessments are conducted in three anatomical locations: the lumbar region (close to the application site), the posterior thigh (segmentally related area), and the forearm (unrelated site). Additionally, blood flow is assessed using color Doppler ultrasound. Additionally, the sensitivity of the aplicaction site will be also evaluated to assess the cream effects.

The study aims to improve understanding of the peripheral mechanisms involved in magnetic tape application, clarify the potential neuromodulatory role of cutaneous afferents, and determine whether the observed effects are mediated through local sensory mechanisms

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults (18-35 years old)
* Participants interested in laser hair removal who have a prior prescription for EMLA cream

Exclusion Criteria:

* Pregnancy
* Severe illnesses: diabetes, cancer, neurological conditions, depression, etc.
* Dermatological conditions or skin alterations (large wounds, scars, or tattoos)
* Allergy to lidocaine or prilocaine (components of EMLA cream)
* Having exercised within the previous 12 hours
* Use of any toxic substances or caffeine intake within the previous 12 hours
* Undergoing laser hair removal in the lumbar, posterior thigh, or anterior forearm areas within the past 24-48 hours

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Mechanical pain sensitivity (300g Von Frey monofilament) | Baseline (pre-intervention), Post-cream (immediately after cream removal), Mid-intervention (with tape on), and Immediate Post-intervention (immediately after tape removal) at each weekly visit (Visits 1-4)
  Pain intensity will be assessed using a 300g Von Frey filament applied to the skin. Participants will report pain on an 11-point verbal Numeric Rating Scale (vNRS) from 0 (no pain) to 10 (worst imaginable pain). This measurement is performed in three regions (lumbar area, posterior thigh, and forearm) before and after each intervention. Higher NRS scores indicate greater mechanical pain sensitivity.
  Additionally, it will be applied on intervention location site to assess the cream effect and confirm the anesthetic effects

SECONDARY OUTCOMES:
Mechanical Detection Threshold (Von Frey Filaments) | Baseline (pre-intervention), Post-cream (immediately after cream removal), Mid-intervention (with tape on), and Immediate Post-intervention (immediately after tape removal) at each weekly visit (Visits 1-4)
  A set of von Frey filaments of increasing thickness (0.008-300 g) will be applied until the participant detects the stimulus in 3 out of 5 attempts. The smallest filament force (in grams) perceived is recorded as the threshold. Measurements are taken in the lumbar region, posterior thigh, and forearm. Higher thresholds indicate reduced tactile sensitivity.
  Additionally, it will be applied on intervention location site to assess the cream effect and confirm the anesthetic effects
Pressure Pain Threshold (Algometer) | Baseline (pre-intervention), Mid-intervention (with tape on) and Immediate Post-intervention (immediately after tape removal) at each weekly visit (Visits 1-4)
  A digital algometer with a 1-cm² probe will be pressed gradually (1 kg/s) against the skin until participants report the first painful sensation. The force (kg/cm²) at which pain is first perceived is the PPT. Measurements are taken twice at each site (lumbar, thigh, forearm), and the average is used for analysis. Higher PPT values indicate lower pain sensitivity
Painful pressure sensitivity (algometer) | Baseline (pre-intervention), Mid-intervention (with tape on) and Immediate Post-intervention (immediately after tape removal) at each weekly visit (Visits 1-4)
  A standard pressure of 5 kg is applied with an algometer on the lumbar region, thigh and forearm. Participants rate their pain on a 0-10 verbal Numeric Rating Scale (vNRS). This is done twice and averaged. Higher scores indicate greater evoked pain under a fixed force
Blood Flow Assessed by Color Doppler Ultrasound | Baseline (pre-intervention), Mid-intervention (5 min with tape on) and Immediate Post-intervention (5 min after tape removal) at each weekly visit (Visits 1-4)
  Blood flow in the paravertebral lumbar region, thigh and forearm will be assessed using power Doppler ultrasound. Perfusion parameters (e.g., number of color signals, fractional moving blood volume) are recorded over 20-30 seconds at rest, before and after the intervention. Higher perfusion values may indicate increased blood flow
Assessment of participant blinding post-intervention | Immediately Post-intervention after each of the four intervention visits (Visits 1-4)
  After each session, participants complete a brief questionnaire indicating whether they believe they received magnetic or placebo tape, and anesthetic or moisturizing cream. The proportion of correct guesses is used to evaluate blinding effectiveness

IPD SHARING:
Plan to Share IPD: Yes
It will shared the IPD used in the results publication
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Smith E, Azzopardi C, Thaker S, Botchu R, Gupta H. Power Doppler in musculoskeletal ultrasound: uses, pitfalls and principles to overcome its shortcomings. J Ultrasound. 2021 Jun;24(2):151-156. doi: 10.1007/s40477-020-00489-0. Epub 2020 Jul 18. PMID 32683646
- [Background] Sillevis R, Cuenca-Zaldivar JN, Fernandez-Carnero S, Garcia-Haba B, Sanchez Romero EA, Selva-Sarzo F. Neuromodulation of the Autonomic Nervous System in Chronic Low Back Pain: A Randomized, Controlled, Crossover Clinical Trial. Biomedicines. 2023 May 26;11(6):1551. doi: 10.3390/biomedicines11061551. PMID 37371646
- [Background] Selva-Sarzo F, Fernandez-Carnero S, Sillevis R, Hernandez-Garces H, Benitez-Martinez JC, Cuenca-Zaldivar JN. The Direct Effect of Magnetic Tape(R) on Pain and Lower-Extremity Blood Flow in Subjects with Low-Back Pain: A Randomized Clinical Trial. Sensors (Basel). 2021 Sep 29;21(19):6517. doi: 10.3390/s21196517. PMID 34640836
- [Background] Rampazo EP, Martignago CCS, de Noronha M, Liebano RE. Transcutaneous electrical stimulation in neck pain: A systematic review and meta-analysis. Eur J Pain. 2022 Jan;26(1):18-42. doi: 10.1002/ejp.1845. Epub 2021 Aug 3. PMID 34288255
- [Background] Popescu A, Lee H. Neck Pain and Lower Back Pain. Med Clin North Am. 2020 Mar;104(2):279-292. doi: 10.1016/j.mcna.2019.11.003. Epub 2019 Dec 20. PMID 32035569
- [Background] Newman JS, Adler RS, Rubin JM. Power Doppler sonography: use in measuring alterations in muscle blood volume after exercise. AJR Am J Roentgenol. 1997 Jun;168(6):1525-30. doi: 10.2214/ajr.168.6.9168718.
- [Background] Lin S, Zhu B, Huang G, Wang C, Zeng Q, Zhang S. Short-Term Effect of Kinesiotaping on Chronic Nonspecific Low Back Pain and Disability: A Meta-Analysis of Randomized Controlled Trials. Phys Ther. 2020 Feb 7;100(2):238-254. doi: 10.1093/ptj/pzz163. PMID 31696916
- [Background] Lall MP, Restrepo E. The Biopsychosocial Model of Low Back Pain and Patient-Centered Outcomes Following Lumbar Fusion. Orthop Nurs. 2017 May/Jun;36(3):213-221. doi: 10.1097/NOR.0000000000000350. PMID 28538537
- [Background] Kolahi J, Bang H, Park J. Towards a proposal for assessment of blinding success in clinical trials: up-to-date review. Community Dent Oral Epidemiol. 2009 Dec;37(6):477-84. doi: 10.1111/j.1600-0528.2009.00494.x. Epub 2009 Sep 15. PMID 19758415
- [Background] Knezevic NN, Candido KD, Vlaeyen JWS, Van Zundert J, Cohen SP. Low back pain. Lancet. 2021 Jul 3;398(10294):78-92. doi: 10.1016/S0140-6736(21)00733-9. Epub 2021 Jun 8. PMID 34115979
- [Background] Kazeminasab S, Nejadghaderi SA, Amiri P, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Neck pain: global epidemiology, trends and risk factors. BMC Musculoskelet Disord. 2022 Jan 3;23(1):26. doi: 10.1186/s12891-021-04957-4. PMID 34980079
- [Background] Heres HM, Schoots T, Tchang BCY, Rutten MCM, Kemps HMC, van de Vosse FN, Lopata RGP. Perfusion dynamics assessment with Power Doppler ultrasound in skeletal muscle during maximal and submaximal cycling exercise. Eur J Appl Physiol. 2018 Jun;118(6):1209-1219. doi: 10.1007/s00421-018-3850-y. Epub 2018 Mar 22. PMID 29569054
- [Background] Hayden JA, Ellis J, Ogilvie R, Malmivaara A, van Tulder MW. Exercise therapy for chronic low back pain. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD009790. doi: 10.1002/14651858.CD009790.pub2. PMID 34580864
- [Background] Dori A, Abbasi H, Zaidman CM. Intramuscular blood flow quantification with power doppler ultrasonography. Muscle Nerve. 2016 Nov;54(5):872-878. doi: 10.1002/mus.25108. Epub 2016 Aug 3. PMID 26994405
- [Background] Dias LV, Cordeiro MA, Schmidt de Sales R, Dos Santos MMBR, Korelo RIG, Vojciechowski AS, de Mace do ACB. Immediate analgesic effect of transcutaneous electrical nerve stimulation (TENS) and interferential current (IFC) on chronic low back pain: Randomised placebo-controlled trial. J Bodyw Mov Ther. 2021 Jul;27:181-190. doi: 10.1016/j.jbmt.2021.03.005. Epub 2021 Mar 18. PMID 34391232
- [Background] Corp N, Mansell G, Stynes S, Wynne-Jones G, Morso L, Hill JC, van der Windt DA. Evidence-based treatment recommendations for neck and low back pain across Europe: A systematic review of guidelines. Eur J Pain. 2021 Feb;25(2):275-295. doi: 10.1002/ejp.1679. Epub 2020 Nov 12. PMID 33064878
- [Background] Bozkurt T, Kilic RT, Yosmaoglu HB. The effect of elastic therapeutic taping and rigid taping on pain, functionality, and tissue temperature in lumbar radiculopathy: a randomized controlled study. Somatosens Mot Res. 2021 Dec;38(4):373-380. doi: 10.1080/08990220.2021.1986381. Epub 2021 Oct 12. PMID 34635000
- [Background] Bevan S. Economic impact of musculoskeletal disorders (MSDs) on work in Europe. Best Pract Res Clin Rheumatol. 2015 Jun;29(3):356-73. doi: 10.1016/j.berh.2015.08.002. Epub 2015 Oct 24. PMID 26612235
- [Background] Benarroch EE. Pain-autonomic interactions. Neurol Sci. 2006 May;27 Suppl 2:S130-3. doi: 10.1007/s10072-006-0587-x. PMID 16688616
- [Background] Beltra P, Ruiz-Del-Portal I, Ortega FJ, Valdesuso R, Delicado-Miralles M, Velasco E. Sensorimotor effects of plasticity-inducing percutaneous peripheral nerve stimulation protocols: a blinded, randomized clinical trial. Eur J Pain. 2022 May;26(5):1039-1055. doi: 10.1002/ejp.1928. Epub 2022 Mar 3. PMID 35191131
- [Background] Alfano AP, Taylor AG, Foresman PA, Dunkl PR, McConnell GG, Conaway MR, Gillies GT. Static magnetic fields for treatment of fibromyalgia: a randomized controlled trial. J Altern Complement Med. 2001 Feb;7(1):53-64. doi: 10.1089/107555301300004538. PMID 11246937